CLINICAL TRIAL: NCT01633697
Title: Study of the Effects of Education on Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Kaminsky, MD, Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-131; 1R34HL113290-01 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: COPD
Keywords: emphysema; chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education-Pranayama (Experimental): Subjects will receive education about COPD with special attention to breathing techniques
  Interventions: Behavioral: Pranayama
- Education-Control (Sham Comparator): Subjects will receive education alone about COPD.
  Interventions: Behavioral: Education alone

INTERVENTIONS:
Behavioral: Pranayama — Specific yoga-related breathing method.
  Other Names: Dirgha 3-Part Breathing method
  Arms: Education-Pranayama
Behavioral: Education alone — No special attention to breathing
  Arms: Education-Control

SUMMARY:
The investigators hypothesize that education will improve exercise capacity, symptoms and quality of life in patients with chronic obstructive pulmonary disease (COPD). In addition, the investigators are interested in determining how education might alter various chemicals in the blood and exhaled breath that reflect inflammation in the lungs and the body as a whole.

The investigators plan to enroll 42 patients into this study, with half of them participating at each of the two sites, Vermont Lung Center at the University of Vermont in Burlington, Vermont, and at Baylor College of Medicine in Houston, Texas. Participants will undergo a series of measurements and tests at the beginning of the study, receive formal education about COPD over the next 2 weeks, return at 6 weeks for a brief refresher session, and finally return after 12 weeks for repeat measurement and testing as was done at the beginning. Participants will be asked to keep a diary of symptoms, medication, and exercise during the study.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major health problem worldwide, and is currently the third leading cause of death in the United Sates. Patients with COPD mainly complain of shortness of breath with daily activities and exercise. A key mechanism of dyspnea is dynamic hyperinflation, or air trapping, which results from the severe airflow limitation that characterizes the disease. Inhaled bronchodilators and corticosteroids may help, but these therapies are expensive and may have side effects. Pulmonary rehabilitation is very effective at reducing dyspnea and improving exercise tolerance, but it is not widely available to patients. The investigators propose studying the effect of a simple breathing exercise known as pranayama, or yogic breathing. The central hypothesis is that the practice of pranayama will improve exercise tolerance in patients with COPD. The investigators believe that the mechanisms involved will include reduced dynamic hyperinflation as well as beneficial effects on lung mechanics, inflammation and oxidative stress. This hypothesis will be tested in a randomized, double blind, controlled trial of pranayama vs. usual care (education) in COPD patients. In Specific Aim 1, the investigators will determine the effect of pranayama on exercise tolerance as measured by 6 min walk distance; in Specific Aim 2, the investigators will determine the effect of pranayama on dynamic hyperinflation as measured by changes in inspiratory capacity before and after exercise; and in Specific Aim 3, The investigators will determine the effect of pranayama on oxidative stress systemic inflammation, shortness of breath, and quality of life. The study is designed to be applicable to a wide variety of clinical settings, since it will involve two diverse clinical sites (Burlington, VT and Houston, TX), require minimal direct intervention, and engage participants in self-learning and practice. The data from this study will provide fundamental new insights into the mechanisms of action of pranayama, and will be critical in designing a large, multicenter trial to test the effectiveness of pranayama in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 and older, with a physician diagnosis of COPD
* COPD defined according to GOLD criteria, with FEV1/FVC < 0.7, and FEV1 < 80% predicted.
* Current non-smoker
* Stable medical regimen for COPD over last 4 weeks
* Stable physical activity over the last 4 weeks, with no plans for any change during the duration of the study
* MRC Dyspnea Scale > 2
* Not planning to engage in any formal pulmonary rehabilitation program during the time of the study
* No use of any nutritional supplements other than standard multivitamins

Exclusion Criteria:

* Exacerbation of disease within previous 2 weeks
* Concomitant other respiratory disease or significant cardiovascular disease
* Previous practice of yoga
* Current use of antioxidant supplements (e.g., vitamin C, vitamin E, n-acetylcysteine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 12 weeks
  Exercise tolerance will be measured by 6 min walk distance at baseline and again after 12 weeks of the intervention

SECONDARY OUTCOMES:
Dynamic hyperinflation | 12 weeks
  Dynamic hyperinflation will be measured by changes in inspiratory capacity that occur before and after the 6 min walk test, at baseline, and then again at 12 weeks.
Oxidative stress | 12 weeks
  Oxidative stress will be measured by levels of H2O2, 8-isoprostane, and glutathione in exhaled breath condensate at baseline and again at 12 weeks.
Systemic inflammation | 12 weeks
  Systemic inflammation will be assessed by plasma levels of CRP, IL-6 and red cell distribution width at baseline and at 12 weeks.
Lung mechanics | 12 weeks
  Lung mechanics will be assessed by measurement of respiratory system impedance using the forced oscillation technique at baseline and at 12 weeks.
Dyspnea | 12 weeks
  Dyspnea will be assessed by questionnaires (Borg, MRC, BDI/TDI) at baseline and at 12 weeks.
Quality of Life | 12 weeks
  Quality of life will be assessed by the St. George Respiratory Questionnaire at baseline and at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David Kaminsky, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center, Colchester, Vermont

REFERENCES:
- See also: Vermont Lung Center — http://www.med.uvm.edu/vermontlung/HP-DEPT.asp?SiteAreaID=513